CLINICAL TRIAL: NCT00628563
Title: REALL STUDY: A Retrospective Observational Study to Compare the Effectiveness and Cost-effectiveness Between Different Step-3 Asthma Treatment Strategies in Real Life Patients in Primary Care
Brief Title: REALL: A Retrospective Observational Study to Compare the Effectiveness and Cost-Effectiveness Between Different Step-3 Asthma Treatment Strategies
Acronym: REALL
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: GP501RGD0685
Record Dates: First submitted 2008-01-31; First posted 2008-03-05 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Asthma patients

SUMMARY:
This is a retrospective observational study utilising anonymised individual patient clinical and prescribing information routinely collected by UK General Practitioners (GPs). This information will be observed for two years, one year pre and one year post- "Index Prescription Date" (IPD). The IPD is the date when a patient was first switched to any option of the step-3 asthma treatment regimen. The one year before the IPD is the baseline period and will be reviewed for risk factors and confounding factors. The one year after the IPD is the outcome period and will be observed to see the outcomes of the new treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a physician diagnosis of asthma who have stepped-up to any option of step-3 asthma treatment (trial therapy), and;
2. Patients with the trial therapy who have data in their records for at least one year for the baseline period and at least one year for the outcome period.

Exclusion Criteria:

1. Patients who were not prescribed with any option of step-3 treatment (the trial therapy) during the study period.
2. Patients treated with the trial therapy, but do not have data in their records for at least one year for the baseline period and at least one year for the outcome period.
3. Patients treated with long-acting anticholinergic drugs, either alone or in combination with other therapy.
4. Patients with a physician diagnosis of COPD with or without asthma.
5. Patients who have resolved from asthma; i.e. patients who were previously diagnosed as having asthma, have now been undiagnosed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with a physician diagnosis of asthma who have stepped-up to any option of step-3 asthma treatment (trial therapy), and;
  2. Patients with the trial therapy who have data in their records for at least one year for the baseline period and at least one year for the outcome period.
Sampling Method: Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 2007-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The achievement of asthma control. This will be assessed by evaluating the patient data for one year in the outcome period. On this basis patients will be divided into two groups | 1 year

SECONDARY OUTCOMES:
The asthma control will be monitored, directly from patients' point of view, by Royal College of Physician (RCP) 3 questions at least after 6 months of IPD (British Thoracic Society (BTS) July, 2007). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Principal Investigator — University of Aberdeen
Locations (1):
- Medical Practices, UK, United Kingdom